CLINICAL TRIAL: NCT01799824
Title: Clinical Trial to Evaluate ANT-1403 in the Treatment of Primary Axillary Hyperhidrosis in Adults
Brief Title: Clinical Trial to Evaluate ANT-1403 in the Treatment of Primary Axillary Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anterios Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANT-1403-HHID-202
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-11

CONDITIONS: Primary Axillary Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): ANT-1403
  Interventions: Biological: ANT-1403
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: ANT-1403
  Arms: Active
Biological: placebo
  Arms: Vehicle

SUMMARY:
The purpose of this study is to confirm the effect of ANT-1403 in the treatment of primary axillary hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 - 70 years of age
* diagnosis of moderate to severe primary axillary hyperhidrosis
* ≥50 mg of sweat production/axilla in 5 minutes as measured gravimetrically
* HDSS score of ≥3

Exclusion Criteria:

* diagnosis of secondary hyperhidrosis
* skin affliction in the axilla requiring medical treatment
* 20% aluminum hydrochloride, e.g. Drysol®, in 2 weeks prior of Baseline
* oral anticholinergic treatment
* botulinum toxin treatment in the prior 9 months
* history of surgery for axillary hyperhidrosis
* present or history of neuromuscular disease
* female subjects who are pregnant or are nursing a child

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
HDSS | Week 8

SECONDARY OUTCOMES:
GSP | Week 8

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Miami, Florida
  - Pinellas Park, Florida
  - West Palm Beach, Florida
  - Louisville, Kentucky
  - East Windsor, New Jersey
  - Rochester, New York
  - Raleigh, North Carolina
  - Yardley, Pennsylvania
  - Norfolk, Virginia